CLINICAL TRIAL: NCT07085702
Title: A Phase 1 Randomized, Placebo-controlled, Observer-blind Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of the GSK 4-component Vaccine Against Group A Streptococcus Pyogenes (Strep A) With Alum or AS37 in Healthy Adults 18 to 25 Years of Age in Australia
Brief Title: A Study to Evaluate Safety, Reactogenicity, and Immunogenicity of the GSK 4-component Strep A Vaccine With Aluminum Hydroxide (Alum) or AS37 in Healthy Young Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: HHS/BARDA (Unknown); Wellcome Trust (Other); DHSC/GAMRIF (Unknown); Germany/BMBF (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 217935; 75A50122C00028 (Other Grant/Funding Number: HHS/BARDA); 224842/Z/21/Z (Other Grant/Funding Number: Wellcome Trust); 2-28-23 (Other Grant/Funding Number: DHSC/GAMRIF)
Record Dates: First submitted 2025-07-11; First posted 2025-07-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Streptococcal Infections
Keywords: Strep A; Streptococcus pyogenes; Safety; Reactogenicity; Immunogenicity; Healthy Adults; Australia
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Observer-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Low dose Strep A Alum Group (Experimental): Participants randomized to receive 3 doses of Low dose Strep A Alum vaccine on Day 1, Day 31, and Day 121.
  Interventions: Biological: Low dose Strep A Alum
- Medium dose Strep A Alum Group (Experimental): Participants randomized to receive 3 doses of Medium dose Strep A Alum vaccine on Day 1, Day 31, and Day 121.
  Interventions: Biological: Medium dose Strep A Alum
- High dose Strep A Alum Group (Experimental): Participants randomized to receive 3 doses of High dose Strep A Alum vaccine on Day 1, Day 31, and Day 121.
  Interventions: Biological: High dose Strep A Alum
- Low dose Strep A AS37 Group (Experimental): Participants randomized to receive 3 doses of Low dose Strep A AS37 vaccine on Day 1, Day 31, and Day 121.
  Interventions: Biological: Low dose Strep A AS37
- Medium dose Strep A AS37 Group (Experimental): Participants randomized to receive 3 doses of Medium dose Strep A AS37 vaccine on Day 1, Day 31, and Day 121.
  Interventions: Biological: Medium dose Strep A AS37
- High dose Strep A AS37 Group (Experimental): Participants randomized to receive 3 doses of High dose Strep A AS37 vaccine on Day 1, Day 31, and Day 121.
  Interventions: Biological: High dose Strep A AS37
- Strep A Alum Placebo Group (Placebo Comparator): Participants randomized to receive 3 doses of Strep A Alum Placebo on Day 1, Day 31, and Day 121.
  Interventions: Drug: Strep A Alum Placebo

INTERVENTIONS:
Biological: Low dose Strep A Alum — Low dose Strep A Alum vaccine will be administered intramuscularly (IM)
  Arms: Low dose Strep A Alum Group
Biological: Medium dose Strep A Alum — Medium dose Strep A Alum vaccine will be administered IM
  Arms: Medium dose Strep A Alum Group
Biological: High dose Strep A Alum — High dose Strep A Alum vaccine will be administered IM
  Arms: High dose Strep A Alum Group
Biological: Low dose Strep A AS37 — Low dose Strep A AS37 vaccine will be administered IM
  Arms: Low dose Strep A AS37 Group
Biological: Medium dose Strep A AS37 — Medium dose Strep A AS37 vaccine will be administered IM
  Arms: Medium dose Strep A AS37 Group
Biological: High dose Strep A AS37 — High dose Strep A AS37 vaccine will be administered IM
  Arms: High dose Strep A AS37 Group
Drug: Strep A Alum Placebo — Strep A Alum Placebo will be administered IM
  Arms: Strep A Alum Placebo Group

SUMMARY:
The purpose of this study is to assess the safety of 3 doses of 2 new Strep A vaccine formulations, one with an Alum adjuvant, and the other with AS37 adjuvant. The Strep A vaccine will be tested for the first time in humans, in healthy young adults 18 to 25 years of age. The study will also assess if the vaccines have any immediate reactions and if they induce an immune response. A low, medium, and high dose of each formulation of the vaccine will be assessed in sequence.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who, in the opinion of the Investigator, can and will comply with the requirements of the protocol (e.g., completion of electronic diaries [eDiaries], return for follow-up visits).
* Written or witnessed/thumb-printed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history, clinical examination, and laboratory assessments.
* Satisfies all screening requirements.
* Male and female participants between and including 18 and 25 years of age at the time of informed consent.
* Female participants of nonchildbearing potential may be enrolled in the study. Nonchildbearing potential is defined as premenarche, postmenopause, or had current bilateral tubal ligation or occlusion, hysterectomy, or bilateral ovariectomy.
* Female participants who are of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire study intervention administration period and for 1 month after completion of the study intervention administration series.
* Male participants who are sexually active with a female partner of childbearing potential are eligible to participate if they agree to have their partner use a highly effective method of contraception for 1 month prior to the first study intervention administration until 1 month after completion of the study intervention administration series.
* Male participants must refrain from donating sperm for 1 month prior to the first study intervention administration until 1 month after completion of the study intervention administration series.
* Participants seronegative for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C at Screening.

Exclusion Criteria:

* History of rheumatic fever or rheumatic heart disease during the lifetime of the participant as confirmed during interview with the participant or as documented in medical records.
* Recent history of pharyngitis in the last four (4) weeks will be excluded. These participants can be rescreened once the recent pharyngitis passes the 4-weeks period. Participants with symptoms of acute pharyngitis at Screening will be tested with a Strep A rapid antigen test. Those with positive results will be excluded.
* Progressive, unstable, or uncontrolled clinical conditions.
* History (known or suspected) of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity (e.g., allergy) to medicinal products or medical equipment anticipated to be used in this study.
* Clinical conditions that represents a contraindication for IM vaccination or blood draws.
* Any behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the participant's ability to participate in the study.
* Acute disease and/or fever (defined as temperature >=38.0°C) at the time of enrollment.
* Any Grade >=2 and/or clinically significant hematological and/or biochemical laboratory abnormality.
* Any echocardiographic/Doppler Echo findings consistent with carditis at Screening.
* Recurrent history or uncontrolled neurological disorders or seizures.
* Medical history or family history of autoimmune disease and other pIMDs.
* Family history of acute rheumatic fever.
* Acute or chronic illness, or clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality.
* Any other clinical condition that might pose additional risk to the participant due to participation in the study.
* Administration of long-acting immune-modifying drugs (e.g., infliximab) at any time prior to the administration of the first dose of study intervention(s) or planned administration during the study period.
* Prior receipt of an experimental Strep A vaccine.
* Use of any investigational or nonregistered product (drug, vaccine, or medical device) other than the study interventions during the period starting 30 days before the first dose of study intervention (Day -30 to Day 1), or their planned use during the study period.
* Receipt of a vaccine not foreseen by the study protocol administered during the period starting at 21 days before the first dose of study intervention (28 days before the first dose, in case of live vaccines) and ending after the last dose of study intervention administration.
* Administration of immunoglobulins and/or any blood products or plasma derivatives, or bone marrow transplantation, during the period starting 3 months before administration of the first dose of study intervention(s) or planned administration during the study period.
* Chronic administration (defined as >14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first dose of study intervention. For corticosteroids, this means prednisone equivalent >=20 mg/day for adult participants. Inhaled, topical, intra-articular, and intranasal steroids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug, vaccine, or invasive medical device).
* Pregnant or lactating female participant.
* Participant who is planning to become pregnant or planning to discontinue contraceptive precautions.
* History of or current chronic alcohol consumption and/or drug abuse.
* Any study personnel or their immediate dependents, family, or household members.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with solicited administration site events | Up to 7 days after each study intervention administration occurring at Day 1, Day 31, and Day 121
  Solicited administration-site events include pain, redness, and swelling at the administration site.
Number of participants with solicited systemic events | Up to 7 days after each study intervention administration occurring at Day 1, Day 31, and Day 121
  Solicited systemic events include fever, headache, myalgia (muscle pain), arthralgia (joint pain), and fatigue (tiredness). Fever is defined as body temperature equal to or above 38.0°C. The preferred location for measuring temperature is the axilla.
Number of participants with unsolicited adverse events (AEs) | Up to 30 days after each study intervention administration occurring at Day 1, Day 31, and Day 121
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs.
Number of participants with laboratory abnormalities | 7 days after each study intervention administration at Day 8, Day 38, and Day 128
Number of participants with adverse events of special interest (AESIs) | From Day 1 to Day 301
  AESIs include potential immune-mediated disorders (pIMDs) and rheumatic carditis.
Number of participants with serious adverse events (SAEs) | From Day 1 to Day 301
  An SAE is defined as any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongs existing hospitalization, results in disability/incapacity, abnormal pregnancy outcomes, or other medically significant events.
Number of participants with AEs leading to withdrawal from the study or to discontinuation of study vaccine | From Day 1 to Day 301

SECONDARY OUTCOMES:
Geometric mean concentrations of immunoglobulin G (IgG) against Streptolysin O (SLO), S. pyogenes Cell Envelope Protease (SpyCEP), S. pyogenes Adhesion and Division protein (SpyAD), and Group A Carbohydrate (GAC), as measured by multiplex immunoassay | Before each study intervention (Day 1, Day 31, and Day 121), 30 days after each study intervention (Day 31, Day 61, and Day 151), and 7 days and 6 months after the third study intervention administration (Days 128 and 301, respectively)
Geometric mean fold increase of IgG against SLO, SpyCEP, SpyAD, and GAC, as measured by multiplex immunoassay | 30 days after each study intervention administration compared to before each study intervention administration (Day 31 versus Day 1, Day 61 versus Day 31, and Day 151 versus Day 121) and to before study intervention administration (Day 1)
Number of participants with greater than or equal to (>=) 2-fold and >=4 fold increase in IgG antibody concentration against SLO, SpyCEP, SpyAD, and GAC, as measured by multiplex immunoassay | 30 days after each study intervention administration (Day 31, Day 61, and Day 151) compared to before study intervention administration (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: King C Cheung, Principal Investigator — Emeritus Research; Juliet Freeborn, Principal Investigator — Emeritus Research
Locations (2):
- Australia (2):
  - GSK Investigational Site, Botany, New South Wales
  - GSK Investigational Site, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf